CLINICAL TRIAL: NCT04855344
Title: Effect of Deep Brain Stimulation Therapy on Intestinal Microbiota in Patients With Parkinson's Disease
Brief Title: Deep Brain Stimulation Therapy and Intestinal Microbiota
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Ling Zhou
Record Dates: First submitted 2021-04-14; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Deep Brain Stimulation; Gastrointestinal Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to observe the changes of intestinal microbiota after deep brain stimulation (DBS) therapy for Parkinson's disease, and explore the role of intestinal microbiota in the neuroprotective effect of DBS.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age;
2. Primary Parkinson's disease diagnosed according to British Brain Bank criteria (Hoehn and Yahr);
3. Deep brain stimulator therapy;
4. Sign the informed consent.

Exclusion Criteria:

1. Use of probiotics or probiotics during the study;
2. Use antibiotics against intestinal bacteria at present or within the last 1 month;
3. With cognitive dysfunction or mental illness;
4. With severe diseases or is not expected to survive for more than a year;
5. A history of gastrointestinal surgery;
6. AIDS patients, hepatitis B/C positive.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease and are expected to undergo DBS therapy
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in gut microbiota | Baseline (Before deep brain stimulation therapy)/3 month after deep brain stimulation therapy
  Analyzed by 16sRNA sequencing of feces
Change in gut microbiota | Baseline (Before deep brain stimulation therapy)/6 month after deep brain stimulation therapy
  Analyzed by 16sRNA sequencing of feces

SECONDARY OUTCOMES:
Change in blood biomarkers of neuroinflammation and alpha-synuclein | Baseline (Before deep brain stimulation therapy)/3 month after deep brain stimulation therapy
  Comparing the changes of blood biomarkers such as neuroinflammation (TNF-alpha, IL-6, LPS) and alpha-synuclein
Change in blood biomarkers of neuroinflammation and alpha-synuclein | Baseline (Before deep brain stimulation therapy)/6 month after deep brain stimulation therapy
  Comparing the changes of blood biomarkers such as neuroinflammation (TNF-alpha, IL-6, LPS) and alpha-synuclein
Frequency of defecation | Baseline (Before deep brain stimulation therapy)/3 month after deep brain stimulation therapy
Frequency of defecation | Baseline (Before deep brain stimulation therapy)/6 month after deep brain stimulation therapy
Dosage of anti-Parkinson's agent | Baseline (Before deep brain stimulation therapy)/3 month after deep brain stimulation therapy
Dosage of anti-Parkinson's agent | Baseline (Before deep brain stimulation therapy)/6 month after deep brain stimulation therapy
Change in the score of Unified Parkinson's Disease Rating Scales | Baseline (Before deep brain stimulation therapy)/3 month after deep brain stimulation therapy
  It is consisted of six scales, each scale is graded on a scale of 5 (0-4), with zero being normal and 4 being severe.
Change in the score of Unified Parkinson's Disease Rating Scales | Baseline (Before deep brain stimulation therapy)/6 month after deep brain stimulation therapy
  It is consisted of six scales, each scale is graded on a scale of 5 (0-4), with zero being normal and 4 being severe.
Parkinson's Disease Quality of Life Questionnaire-39 (PDQ-39) | Baseline (Before deep brain stimulation therapy)/3 month after deep brain stimulation therapy
  Change in PDQ-39 scores, higher scores mean a worse outcome
Parkinson's Disease Quality of Life Questionnaire-39 (PDQ-39) | Baseline (Before deep brain stimulation therapy)/6 month after deep brain stimulation therapy
  Change in PDQ-39 scores, higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Cunming Liu, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the Hospital Research Ethics Committee of the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China